CLINICAL TRIAL: NCT01775345
Title: Assessment of Different Treatments of Muscle Strengthening in Post-meniscectomy Knee.
Brief Title: Assessment of Different Rehabilitation Treatments After a Partial Removal of the Meniscus
Acronym: MENFIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Principal Investigator, M. Rosa Nogués, University Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MENFIS
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Rehabilitation Post-meniscectomy
Keywords: Partial meniscectomy; Physiotherapy; Isokinetics; Cost-effectiveness
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isotonic exercises + ST (Experimental): This group will realize 20 sessions of muscular force work by means of isotonic exercises, that to the beginning will consist of 2 series of 10 repetitions to 60, 65 and 70 % of a maximum repetition (MR)(MR is the maximum resistance that a muscle can conquer).
  Later, a gradual progression will be realized and the load will be increasing up to being able to realize, before the session 30: 2 series of 15 repetitions to 60, 65 and 70 %, of 1MR, 2 series of 10 repetitions to 75 and 80 % of 1MR and one series of 6 repetitions to 85 and 90 % of 1MR.
  Interventions: Procedure: Isotonic exercises; Procedure: ST
- Isokinetic exercises + ST (Experimental): This group will realize 20 sessions of muscular force work by means of isokinetic exercises, that to the beginning will consist of 2 series of 10 repetitions to 150, 180 and 210 º / seg in the first session and it will be increasing in a progressive and gradual way up to being able to realize, before the last session: 3 series of 15 repetitions to 180 º, 210 º and 240 º / seg, 2 series of 10 repetitions to 120 º and 150 º / seg and 2 series of 6 repetitions of 60 º and 90 º / seg.
  Interventions: Procedure: Isokinetic exercises; Procedure: ST
- Isotonic and isokinetic exercises + ST (Experimental): This group will realize 20 sessions of muscular force work by means of isotonic and isokinetic exercises. To the beginning it will consist of 1 series of 10 repetitions to 150, 180 and 210 º / seg and 1 series of 10 repetitions to 60, 65 and 70 % of 1MR. A gradual progression will be realized up to reaching, before the last session, a load of: 2 series of 15 repetitions to 180, 210 and 240 º / seg, 1 series from 10 to 120 and 150 º / seg and 1 series of 6 repetitions to 60 and 90 º / seg, and 1 series of 15 repetitions to 60, 65 and 70 %, of 1MR, 1 series of 10 repetitions to 75 and 80 % of 1MR and 1 series of 3 repetitions to 85 and 90 % of 1MR.
  Interventions: Procedure: Isotonic and isokinetic exercises; Procedure: ST

INTERVENTIONS:
Procedure: Isotonic exercises — 20 sessions of muscular force work by means of isotonic exercises, that to the beginning will consist of 2 series of 10 repetitions to 60, 65 and 70 % of a MR.
  Later, a gradual progression will be realized and the load will be increasing up to being able to realize, before the session 30: 2 series of 15 repetitions to 60, 65 and 70 %, of 1MR, 2 series of 10 repetitions to 75 and 80 % of 1MR and one series of 6 repetitions to 85 and 90 % of 1MR.
  Arms: Isotonic exercises + ST
Procedure: Isokinetic exercises — 20 sessions of muscular force work by means of isokinetic exercises, that to the beginning will consist of 2 series of 10 repetitions to 150, 180 and 210 º / seg in the first session and it will be increasing in a progressive and gradual way up to being able to realize, before the last session: 3 series of 15 repetitions to 180 º, 210 º and 240 º / seg, 2 series of 10 repetitions to 120 º and 150 º / seg and 2 series of 6 repetitions of 60 º and 90 º / seg.
  Arms: Isokinetic exercises + ST
Procedure: Isotonic and isokinetic exercises — 20 sessions of muscular force work by means of isotonic and isokinetic exercises. To the beginning it will consist of 1 series of 10 repetitions to 150, 180 and 210 º / seg and 1 series of 10 repetitions to 60, 65 and 70 % of 1 MR. A gradual progression will be realized up to reaching, before the last session, a load of: 2 series of 15 repetitions to 180, 210 and 240 º / seg, 1 series from 10 to 120 and 150 º / seg and 1 series of 6 repetitions to 60 and 90 º / seg, and 1 series of 15 repetitions to 60, 65 and 70 %, of 1MR, 1 series of 10 repetitions to 75 and 80 % of 1MR and 1 series of 3 repetitions to 85 and 90 % of 1MR.
  Arms: Isotonic and isokinetic exercises + ST
Procedure: ST — Standard therapy: The 10 first rehabilitation sessions will be common (manual therapy, electrotherapy, proprioceptive reeducation, isometric exercises, bike exercise and cryotherapy)
  Other Names: Standard therapy

SUMMARY:
To determine that rehabilitation treatment for a partial meniscectomy is more efficient in the functional recovery of the knee. Set in the fewest possible sessions, what treatment has benefits that last beyond the physical and what is the best cost-effectiveness.

It is expected that the combination of isotonic and isokinetic exercises in post-meniscectomy physiotherapy allows faster and less costly patient rehabilitate than the current isotonic protocol.

DETAILED DESCRIPTION:
Longitudinal randomized single-blind study, 81 patients (27 per group; 3 groups), 18 to 60 years, underwent surgery meniscus and performing rehabilitation at the University Hospital Sant Joan de Reus. The first rehabilitation sessions will be common (manual therapy, electrotherapy, proprioceptive reeducation, isometric exercises, bike exercise and cryotherapy). From Session 10, will be randomized into 3 groups: group 1 protocol added isotonic exercises, group 2 isokinetic exercises and group 3 isotonic and isokinetic exercises.

The principal variable will be the maximum force peak of the muscle. An evaluation of other parameters such as knee function (Lysholm Test) and the degree of pain (VAS) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of between 18 and 60 years
* Surgical Intervention: partial meniscectomy of the internal meniscus
* Informed consent

Exclusion Criteria:

* Re-meniscectomy
* Associate injury of crossed ligaments
* Degenerative osteoarthritis of knee degree the II, III or IV
* Morbid obesity
* Infectious diseases in the skin, cutaneous injuries and / or zones of hypoesthesia
* Participants with malignant tumors
* Participants with cognitive or sensory alterations
* Volunteers who have taken part in a study in the last 3 months
* Lack of collaboration of the patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maximum force peak in flexion of 60 º / seg and 180 º / seg, and extension of 60 º / seg and 180 º / seg. The assessment will be comparative. It will be realized in both the affected knee and the healthy knee. | 7 weeks
  We will observe the maximum force peak in flexion of 60 º / seg and 180 º / seg, and extension of 60 º / seg and 180 º / seg. Both the valuation and the work of muscular involution with isokinetic exercises will fulfil with an isokinetic dynamometer Biodex 3.

SECONDARY OUTCOMES:
Knee functionality with the Lysholm Test. | 7 weeks
  Questionnaire with 8 questions that the patient must answer with regard to the functionality of the affected knee. Maximum functionality 100 points.

OTHER OUTCOMES:
Degree of pain with the Visual Analogue Scale (VAS). | 7 weeks
  The patients must mark, in a scale from 0 to 10, the pain that they perceive in the affected knee, being 10 the maximum possible pain.
Metabolomic biomarkers | 7 weeks
  To identify changes in the metabolomic biomarkers related to inflammation process along the study, 3 plasma samples will be collected from patients: one week before the day of the surgical procedure, the 1st day of rehabilitation programme and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Casajuana, PT, Study Director — Hospital Universitari Sant Joan de Reus
Locations (1):
- Hospital Universitari Sant Joan, Reus, Spain